CLINICAL TRIAL: NCT05809583
Title: Applying Precision Medicine to Define Predictors of Response to Ozanimod and Discovering Biomarkers in the Management of Ulcerative Colitis Using 7,000 Protein SOMAscan
Brief Title: Define Predictors of Response to Ozanimod in UC Discovering Biomarkers in the Management of Ulcerative Colitis
Status: Withdrawn | Type: Observational
Why Stopped: Funding withdrawn
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Laurie Grossberg, Instructor in Medicine, Beth Israel Deaconess Medical Center
Other Study IDs: 2022P000954
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Ulcerative Colitis
Keywords: biomarkers; ozanimod; somascan
MeSH Terms: conditions — Colitis, Ulcerative | interventions — ozanimod

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ozanimod: Patients with UC starting ozanimod therapy as part of their clinical care
  Interventions: Drug: Ozanimod

INTERVENTIONS:
Drug: Ozanimod — Patients with established diagnosis of UC starting ozanimod therapy as part of their clinical care

SUMMARY:
A diagnostic tool that identifies biomarkers that predict response prior to and during induction of ozanimod will have a major impact on improving outcomes in UC patients. Using SOMAscan from SomaLogic (Boulder, CO), our study aims to discover serum protein biomarkers in UC patients that predict response to ozanimod and to gain insight into the pathophysiological mechanisms underlying ozanimod response.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years of age with established diagnosis of UC starting ozanimod therapy as part of their clinical care
2. Patients with moderate to severe UC, determined by a 3-component Mayo score of 5-9 with an endoscopic subscore ≥ 2.Endoscopy must be performed within 90 days of ozanimod initiation
3. Elevated CRP (greater than upper limit of normal on assay) and/or fecal calprotectin (>250 mcg/g) within 90 days of drug initiation

Exclusion Criteria:

1. Diagnosis of Crohn's disease or indeterminate colitis
2. Total (procto)colectomy
3. Ileoanal pouch anastomosis
4. Current ileostomy or colostomy
5. Untreated Clostridium difficile infection
6. Known pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients ≥18 years of age with established diagnosis of UC starting ozanimod therapy as part of their clinical care
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Clinical response | 10 weeks
  The primary endpoint measure is clinical response defined as a decrease of at least 50% in PRO2 at week 10 (end of induction)

SECONDARY OUTCOMES:
Clinical response | 22 weeks
  Clinical response defined as a decrease of at least 50% in PRO2 at week 22
Clinical remission | 10 weeks
  Symptomatic/PRO2 remission defined as stool frequency subscore of 0 or 1 and rectal bleeding subscore of 0 at weeks 10 and 22.
Fecal calprotectin | 2, 10, 22 weeks
  Change from baseline in level of fecal calprotectin at weeks 2, 10, and 22
CRP | 2, 10, 22 weeks
  Change from baseline in level of CRP at weeks 2, 10, 22
Corticosteroid free remission | 22 weeks
  Corticosteroid free remission at week 22

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Grossberg, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No